CLINICAL TRIAL: NCT06003998
Title: Intraperitoneal Irinotecan With Concomitant FOLFOX and Bevacizumab for Patients With Unresectable Colorectal Peritoneal Metastases
Brief Title: Intraperitoneal Irinotecan With Concomitant FOLFOX and Bevacizumab
Acronym: INTERACT-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, J. W. A. Burger, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL81672.100.22
Record Dates: First submitted 2022-11-08; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
Keywords: Peritoneal metastases; colorectal cancer; Intraperitoneal; Irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Folfox protocol; Fluorouracil; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal irinotecan 75 mg + mFOLFOX-4 and bevacizumab (Experimental): Intraperitoneal irinotecan, 75 mg flat dose + systemic oxaliplatin, 5-Fluorouracil and bevacizumab (mFOLFOX+beva) (dose via standard of care)
  Interventions: Drug: Irinotecan; Drug: FOLFOX regimen; Drug: Bevacizumab

INTERVENTIONS:
Drug: Irinotecan — 2 weekly IP irinotecan (max 12 cycles), dose 75 mg flat dose
  Other Names: Intraperitoneal irinotecan
Drug: FOLFOX regimen — FOLFOX-4 regimens consist of 85 mg/m2 oxaliplatin plus 200 mg/m2 LV and 5-FU 400 mg/m2 bolus on day 1 followed by 1600 mg/m2 5-FU as a 46-h infusion
  Other Names: 5-FU + oxaliplatin
Drug: Bevacizumab — Bevacizumab according to standard of care
  Other Names: Avastin

SUMMARY:
The rationale of the current study is that the addition of intraperitoneal irinotecan (75 mg) to palliative systemic therapy is feasible and safe, and might result in an increased overall and progression free survival in patients with unresectable colorectal peritoneal metastases. The primary objectives are to explore the overall survival for the addition of intraperitoneal irinotecan (75 mg) to palliative systemic therapy in patients with unresectable colorectal peritoneal metastases. Secondary objectives are to assess the progression-free survival, toxicity profile, patient reported outcomes, costs, tumor response during trial treatment, and the systemic and intraperitoneal pharmacokinetics of irinotecan and SN-38. This is a single-arm, open-label, phase II study and patients will receive intraperitoneal irinotecan (75 mg) in combination with modified FOLFOX4 + bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer;
* Radiologically and clinically or pathologically confirmed unresectable colorectal peritoneal metastases (e.g. PCI >20, extensive small bowel involvement, unresectable disease due to anatomical location);
* WHO performance score of 0-1 with a life expectancy of >3 months;
* Aged 18 years or older;
* Written informed consent;

Exclusion Criteria:

* Presence of extensive systemic metastases that are deemed to be the dominant factor determining prognosis in terms of life expectancy and performance status [e.g. no imminent threat of impaired organ functioning due to the presence of systemic metastases]);
* Prior cytoreductive surgery;
* Prior palliative systemic therapy for colorectal cancer;
* Prior neo-adjuvant/adjuvant systemic therapy for colorectal cancer within the last 6 months;
* Homozygous UGT1A1*28 genotype;
* Homozygous dihydropyrimidine dehydrogenase (DPD) deficiency
* Microsatellite instable (MSI) primary tumor
* Any contra-indication for the planned chemotherapy (e.g. active infection, serious concomitant disease, severe allergy), as determined by the medical oncologist;
* Inadequate organ functions, defined as an haemoglobin of <5 mmol/L, an absolute neutrophil count of <1.5 x 109/L, platelet count of <100 x 109/L, serum creatinine of >1.5 x ULN, creatinine clearance of <30 ml/min, Bilirubin > 2x ULN and liver transaminases of >5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 year
  calculated from (a) the interval from diagnosis of peritoneal metastases until death or last follow-up; (b) the interval from the first day of the first cycle until death or last follow-up).

SECONDARY OUTCOMES:
Progression-free survival | 3 year
  calculated from the interval from the start of trial treatment until first evidence of intraperitoneal and/or systemic disease progression, and/or start of second-line systemic therapy, or last follow-up
Toxicity in CTCAE grading | 28 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Toxicity measured up to four weeks after last cycle.
  Defined as the number of patients who experience / the total number of Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) grade 3-5 adverse events, measured up to four weeks after the last cycle of intraperitoneal irinotecan (75 mg) with concomitant palliative systemic therapy. With the exception of peripheral neuropathy, which will be reported indefinitely, ranging from CTCAE grade 1-5.
Patient-reported outcomes (PROs) with EQ-5D-5L | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Measured one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle.
  Assessed with the 5-level EQ-5D by EuroQol group (EQ-5D-5L) at baseline, one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Patient-reported outcomes (PROs) with EORTC QLQ-C30 | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Measured one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle.
  Assessed with the European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (EORTC QLQ-C30) at baseline, one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle. The EORTC QLQ-C30 comprises 30 items, 24 of which are aggregated into nine multi-item scales, that is, five functioning scales, three symptom scales and one global health status scale. The remaining six single-item assess symptoms. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Patient-reported outcomes (PROs) with EORTC QLQ-CR29 | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Measured one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle.
  Assessed with the European Organization for Research and Treatment for Cancer Quality of Life Questionnaire, specifically for colorectal cancer (EORTC QLQ-CR29) at baseline, one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle. The resulting QLQ-CR29 consisted of four scales and 19 individual items. Higher scores indicate a higher level of symptoms (i.e. a worse state of the patient).
Healthcare costs | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Measured one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle.
  According to the Dutch manual for cost analysis in health care research, and assessed with the iMTA Medical Consumption Questionnaire at baseline, one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle. The volumes of used healthcare costs were multiplied with the unit costs of these corresponding services.
Productivity loss costs. | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Measured one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle.
  Assessed with the iMTA Productivity Cost Questionnaire at baseline, one week after the first cycle, one week after the fourth cycle, one week after the eighth cycle, and one week after the twelfth cycle.
Occurrence and degree of nephrotoxicity | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles.
  Assessed during standard-of-care laboratory assessment for nephrotoxicity (creatinine, eGFR, and ureum) analysis before each subsequent cycle and graded according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Occurrence and degree of hepatotoxicity | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles.
  Assessed during standard-of-care laboratory assessment for hepatotoxicity (albumin, bilirubin, AST, ALT, LD, AF, yGT) analysis before each subsequent cycle and graded according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Occurrence and degree of haematological toxicity | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles.
  Assessed during standard-of-care laboratory assessment for haematological toxicity (haemoglobin, leucocytes, thrombocyte) analysis before each subsequent cycle and graded according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Response of Tumor marker during treatment | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles.
  Assessed by carcino-embryonic antigen (CEA) analysis during standard laboratory analysis before each subsequent cycle
Number of patients that completed twelve cycles | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles.
  To determine the number of patients completing twelve cycles of treatment with intraperitoneal irinotecan (75 mg) and concomitant palliative systemic therapy, required dose reductions, and reasons for discontinuation.
Objective radiological response | 24 weeks. Each cycle is 2 weeks, maximum of 12 cycles. Measured at baseline, after the fourth cycle, after the eighth cycle, and after the twelfth cycle.
  assessed by thoracoabdominal CT at baseline, after the fourth cycle, after the eighth cycle, and after the twelfth cycle according to RECIST.
Peritoneum/plasma ratio of intraperitoneal irinotecan | 8 weeks. Each cycles is 2 weeks. Measured during cycle 1 and cycle 4.
  To determine the the peritoneum/plasma ratio of intraperitoneal during the first and fourth cycle of intraperitoneal irinotecan (75 mg) and concomitant palliative systemic therapy. Whole blood and peritoneal fluid will be drawn from a peripheral intravenous access and the peritoneal access port, respectively, and collected in 3 mL lithium heparin tubes and 2 mL cryotubes, respectively, at the following moments after the start of irinotecan infusion; t=0, at the end of infusion (EOI), t=30 minutes after EOI and t =2 hrs after EOI and t = 4hrs after EOI. The ratio between the Area Under the Curve (AUC) between irinotecan measured in the peritoneum and measured in the plasma is taken.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - Erasmus Medical Centre, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van de Vlasakker VCJ, Guchelaar NAD, van den Heuvel TBM, Lurvink RJ, van Meerten E, Bax RJF, Creemers GM, van Hellemond IEG, Brandt-Kerkhof ARM, Madsen EVE, Nederend J, Koolen SLW, Nienhuijs SW, Kranenburg O, de Hingh IHJT, Verhoef C, Mathijssen RHJ, Burger JWA; Dutch Peritoneal Oncology Group; Dutch Colorectal Cancer Group. Intraperitoneal irinotecan with concomitant FOLFOX and bevacizumab for patients with unresectable colorectal peritoneal metastases: protocol of the multicentre, open-label, phase II, INTERACT-II trial. BMJ Open. 2024 Jan 18;14(1):e077667. doi: 10.1136/bmjopen-2023-077667. PMID 38238055